CLINICAL TRIAL: NCT07052253
Title: An Open-label, Multicenter, Phase II Clinical Study of AK104/AK112 in Combination With TT-00420 Tablet in Patients With Advanced Hepatocellular Carcinoma.
Brief Title: A Phase II Clinical Study of AK104/AK112 in Combination With TT-00420 Tablet for Advanced HCC.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-223
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1（Safety Lead-In Phase） (Experimental): AK104 10mg/kg Q3W+TT-00420 10mg PO QD （n=3-6）
  Interventions: Drug: TT-00420 (tinengotinib); Drug: AK104
- Cohort 2（Safety Lead-In Phase） (Experimental): AK112 20mg/kg Q3W + TT-00420 10mg PO QD（n=3-6）
  Interventions: Drug: TT-00420 (tinengotinib); Drug: AK112
- Cohort A（Expansion Cohort Phase） (Experimental): AK104 10mg/kg Q3W + TT-00420 10mg PO QD（n=20-30）
  Interventions: Drug: TT-00420 (tinengotinib); Drug: AK104
- Cohort B（Expansion Cohort Phase） (Experimental): AK112 20mg/kg Q3W + TT-00420 10mg PO QD（n=20-30）
  Interventions: Drug: TT-00420 (tinengotinib); Drug: AK112
- Cohort C（Expansion Cohort Phase） (Experimental): TT-00420 10mg PO QD（n=20-30）
  Interventions: Drug: TT-00420 (tinengotinib)

INTERVENTIONS:
Drug: TT-00420 (tinengotinib) — oral
Drug: AK104 — intravenous
  Arms: Cohort 1（Safety Lead-In Phase）; Cohort A（Expansion Cohort Phase）
Drug: AK112 — intravenous
  Arms: Cohort 2（Safety Lead-In Phase）; Cohort B（Expansion Cohort Phase）

SUMMARY:
An Open-label, Multicenter, Phase II Clinical Study of AK104/AK112 in Combination with TT-00420 Tablet in Patients with Advanced Hepatocellular Carcinoma(HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Histologically or cytologically confirmed hepatocellular carcinoma, or meets the clinical diagnostic criteria for hepatocellular carcinoma.
3. Barcelona Clinic Liver Cancer (BCLC) stage C; or stage B and assessed by the investigator as unsuitable for curative topical treatment.
4. For cohorts A and B: No prior systemic anti-cancer treatment for hepatocellular carcinoma.
5. At least one measurable lesion according to RECIST v1.1 criteria.
6. Child-Pugh liver function score ≤7. ECOG performance status of 0 or 1.
7. Clinically controllable HBV or HCV infection.
8. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Previous histologically or cytologically confirmed fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.
2. Diagnosed with another malignancy within 3 years.
3. History of hepatic encephalopathy.
4. Presence of clinically significant pericardial effusion; symptomatic pleural effusion requiring drainage or moderate to severe ascites uncontrolled by diuretics.
5. Concurrent infection with HBV and HCV.
6. Presence of central nervous system metastases or meningeal metastases.
7. Esophageal or gastric variceal bleeding within 6 months. Imaging (CT or MRI) shows extrahepatic metastasis invading major blood vessels or indistinct vascular boundaries, with high bleeding risk assessed by the researcher.
8. Liver tumor volume exceeding 50% of total liver volume; portal vein main trunk tumor thrombus or tumor thrombus in contralateral main branch of the portal vein, or mesenteric vein tumor thrombus; presence of inferior vena cava thrombus or involvement of the heart.
9. Received topical treatment for liver cancer, any systemic anti-tumor drugs, or other clinical trial drugs within 4 weeks prior to the first administration.
10. Unable to swallow, or has severe gastrointestinal disease or gastrointestinal dysfunction. History of intestinal obstruction or intestinal perforation within 6 months.
11. Uncontrolled hypertension, symptomatic heart failure, symptomatic or poorly controlled arrhythmia, myocarditis, cardiomyopathy, history of malignant arrhythmias.
12. Participants with severe bleeding tendencies or coagulation disorders.
13. Active pulmonary tuberculosis, active syphilis, or history of HIV infection.
14. Severe infection within 4 weeks prior to the first administration, or received systemic anti-infective treatment within 14 days.
15. Other conditions with high medical risk or secondary tumor symptoms, which, in the judgment of the researcher, make the participant unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-05-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  assessed by investigator per RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  assessed by investigator per RECIST v1.1
Disease control rate(DCR) | Up to 2 years
  assessed by investigator per RECIST v1.1
Duration of Response (DOR) | Up to 2 years
  assessed by investigator per RECIST v1.1
Time to Response (TTR) | Up to 2 years
  assessed by investigator per RECIST v1.1
Time to Progression (TTP) | Up to 2 years
  assessed by investigator per RECIST v1.1
Overall Survival(OS) | Up to 2 years
  OS is defined as the time from randomization or first dosing to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science And Technology, Wuhan, China